CLINICAL TRIAL: NCT06519162
Title: Exploration of Liver-gut Axis Through Identification of Liver Disease-specific Microbiome
Brief Title: Liver-gut Axis Study Through Identification of Liver Disease-specific Microbiome
Acronym: LGAS
Status: Recruiting | Type: Observational
Sponsor: Chungnam National University Hospital (Other)
Collaborators: Chungnam National University (Other)
Responsible Party: Principal Investigator, HyukSooEun, Associate Professor of Gastroenterology, Chungnam National University Hospital
Other Study IDs: 2024-05-009
Record Dates: First submitted 2024-07-11; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Autoimmune Hepatitis; Primary Sclerosing Cholangitis; Non-Alcoholic Fatty Liver Disease; Liver Abscess; Primary Biliary Cirrhosis
Keywords: Liver Diseases; Microbiota; Immune System
MeSH Terms: conditions — Hepatitis, Autoimmune; Cholangitis, Sclerosing; Non-alcoholic Fatty Liver Disease; Liver Abscess; Liver Cirrhosis, Biliary; Liver Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous whole blood and or Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, we aim to identify gut microbiomes specific to patients with chronic refractory liver disease and to conduct a gut-liver axis study on the pathogenesis and disease progression.

DETAILED DESCRIPTION:
1. The investigators will recruit study participants aged 19 and older who have been diagnosed with autoimmune hepatitis, primary biliary cholangitis, primary sclerosing cholangitis, non-alcoholic steatohepatitis, or liver abscess, along with their household members, and who have agreed to participate in this study at Chungnam National University Hospital.
2. The investigators collect and analyze blood and stool samples from the patients and their household members
3. Sampling Method: Non-Probability Samples
4. Study Population:

Group of autoimmune hepatitis: patients with definite autoimmune hepatitis or their healthy households for controls Group of primary biliary cholangitis: patients with definite primary biliary cholangitis or their healthy households for controls Group of primary sclerosing cholangitis: patients with definite primary sclerosing cholangitis or their healthy households for controls Group of non-alcoholic steatohepatitis: patients with definite non-alcoholic steatohepatitis or their healthy households for controls Group of liver abscess: patients with definite liver abscess or their healthy households for controls.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years and older diagnosed with autoimmune hepatitis, primary biliary cholangitis, primary sclerosing cholangitis, non-alcoholic fatty liver disease, or liver abscess, who have consented to participate in this study at Chungnam National University Hospital.
* Adults aged 19 years and older, who are cohabitants of patients diagnosed with autoimmune hepatitis, primary biliary cholangitis, primary sclerosing cholangitis, non-alcoholic fatty liver disease, or liver abscess, and have consented to participate in this study at Chungnam National University Hospital.

B. Exclusion

Exclusion Criteria:

* Individuals under the age of 19.
* Patients or guardians who do not consent to participate in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients( Autoimmune liver diseases (Autoimmune hepatitis, Primary biliary cholangitis, Primary sclerosing cholangitis), Metabolic liver diseases (Non-alcoholic fatty liver disease) Infectious liver diseases (Liver abscess)
  - their cohabitant
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2029-07-08 (Estimated); Study Completion 2029-07-08 (Estimated)

PRIMARY OUTCOMES:
Chi-square test | Before treatment, 3~12months after treatment
  Using the Galaxy platform, perform taxonomic profiling followed by LDA(Linear Discriminant Analysis ) analysis. Group by primary diagnosis and derive the LDA(Linear Discriminant Analysis) Effect Size, or utilize MaAsLin2(Microbiome Multivariable Association with Linear Models 2) to identify genera/species showing significant compositional changes between diseases.
t-test | Before treatment, 3~12months after treatment
  Using the Galaxy platform, perform taxonomic profiling followed by LDA(Linear Discriminant Analysis) analysis. Group by primary diagnosis and derive the LDA(Linear Discriminant Analysis) Effect Size, or utilize MaAsLin2(Microbiome Multivariable Association with Linear Models 2) to identify genera/species showing significant compositional changes between diseases.
Pearson's coefficient | Before treatment, 3~12months after treatment
  Using the Galaxy platform, perform taxonomic profiling followed by LDA(Linear Discriminant Analysis) analysis. Group by primary diagnosis and derive the LDA(Linear Discriminant Analysis) Effect Size, or utilize MaAsLin2(Microbiome Multivariable Association with Linear Models 2) to identify genera/species showing significant compositional changes between diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Hyuksoo Eun, Principal Investigator — Chungnam National University Hospital
Locations (1):
- Chungnam National University Hospita, Daejeon, Jung-gu, South Korea

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT06519162/Prot_ICF_000.pdf